CLINICAL TRIAL: NCT07060989
Title: A Phase 1/2a Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of NTS071 in Subjects With Advanced Solid Tumors Harboring a TP53 Y220C Mutation
Brief Title: A Study of Safety, Tolerability and Preliminary Efficacy of NTS071 in Subjects With Advanced Solid Tumors Harboring a TP53 Y220C Mutation
Acronym: NTS071
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nutshell Therapeutics (Shanghai) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTS071-101
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; TP53 Y220C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NTS071 (Experimental): Single arm
  Interventions: Drug: NTS071

INTERVENTIONS:
Drug: NTS071 — Oral administration

SUMMARY:
This study is to evaluate the safety, tolerability, PK, and preliminary efficacy of NTS071 in adults with TP53 Y220C-mutated solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2a, first-in-human, open-label, multi-center study with the aim of exploring the safety, tolerability, PK, and preliminary efficacy of NTS071 in subjects with unresectable locally advanced or metastatic solid tumors containing a TP53 Y220C mutation.

This study includes two parts: Phases 1 and 2a. The Phase 1 part consists of the dose escalation and backfill part; The Phase 2a part consists of the cohort expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥ 18 years
2. Advanced solid tumors with TP53 Y220C mutation
3. Previously treated with one or more lines of anticancer therapy and progressive disease
4. At least one measurable lesion according to RECIST version 1.1 criteria
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
6. Adequate organ and bone marrow function

Exclusion Criteria:

1. Known CNS primary tumor and active or untreated CNS metastases
2. History of another primary malignancy that has been diagnosed or required therapy within the past 2 years
3. Toxicities of prior therapy have not been resolved to ≤ Grade 1 or to baseline
4. Significant cardiovascular disease, including congestive heart failure
5. Known hepatitis B, hepatitis C, or human immunodeficiency virus infection that is active
6. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of dose-limiting toxicity (DLT) | The first 26 days of treatment (Cycle 1) per patient
  Incidence of dose-limiting toxicity (DLT) events
Phase 1: incidence of adverse events (AE), serious adverse events (SAEs) | up to 30 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0
Phase 2a: Overall Response Rate (ORR) | Up to 3 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) by Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Phase 1/2a: area under the curve (AUC) | Up to 2 years
  PK parameters to be evaluated for NST071 including area under the curve (AUC) will be determined when appropriate.
Phase 1/2a: maximum concentration (Cmax) | Up to 2 years
  PK parameters to be evaluated for NTS071 including maximum concentration (Cmax) will be determined when appropriate.
Phase 1/2a: half-life (t1/2) of NTS071 | Up to 2 years
  PK parameters to be evaluated for NTS071 including half-life (t1/2) will be determined when appropriate.
Phase 1/2a: trough observed concentrations (Ctrough/Ctau) | Up to 2 years
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of NTS071
Phase 1: Objective response rate (ORR) | Up to 3 years
  To evaluate the preliminary antitumor activity of NTS071
Phase 1/2a: duration of response (DoR) | Up to 3 years
  To evaluate the preliminary anti-tumor activity of NTS071
Phase 1/2a: disease control rate (DCR) | Up to 3 years
  To evaluate the preliminary antitumor activity of NTS071
Phase 1/2a: progression-free survival (PFS) | Up to 3 years
  To evaluate the preliminary antitumor activity of NTS071
Phase 1/2a: Overall survival (OS) | Up to 3 years
  To evaluate the preliminary antitumor activity of NTS071

CONTACTS AND LOCATIONS:
Locations (2):
- Next Oncology, San Antonio, Texas, United States
- Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No